CLINICAL TRIAL: NCT06277765
Title: A Randomized, Double Blind, Placebo-controlled Phase 3 Study to Evaluate the Efficacy and Safety of CM310 in Adolescent Patients With Moderate-to-severe Atopic Dermatitis
Brief Title: Study of CM310 Injection in Adolescent Subjects With Atopic Dermatis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM310-101212
Record Dates: First submitted 2024-02-18; First posted 2024-02-26 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CM310 group (Experimental)
  Interventions: Biological: CM310
- Placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Biological: CM310 — Interleukin-4 receptor(IL-4Rα) monoclonal antibody
  Arms: CM310 group
Other: placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double blind, placebo-controlled phase 3 study to evaluate the efficacy, safety, pharmacokinetics(PK), pharmacodynamics(PD) and immunogenicity of CM310 in children patients with moderate-to-severe atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Have the ability to understand the study and voluntarily sign a written informed consent form (ICF).
* With Atopic Dermatitis.

Exclusion Criteria:

* Not enough washing-out period for previous therapies.
* Any major surgery planned during the research period.
* With intestinal parasitic infection within the 6 months before screening.
* With any circumstance that is not suitable to participate in this study.
* Major surgeries are planned during the study period.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Actual)
Dates: Start 2024-03-21 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving EASI-75 at week 18 | Up to week 18
  The EASI is a composite index with scores ranging from 0 to 72. Four AD disease characteristics (erythema, edema/papulation, excoriation, lichenification) will each be assessed for severity by the investigator on a scale of "0" (none) through "3" (severe).
Proportion of subjects with IGA score of 0 or 1 and a reduction of IGA score by ≥2 points from baseline | up to week 18
  Proportion of subjects with Investigator's Global Assessment (IGA) score of 0 or 1 and a reduction of IGA score by ≥2 points from baseline at week 18. IGA is an assessment instrument used in clinical studies to rate the severity of AD globally, based on a 5-point scale ranging from 0 (clear) to 4 (severe).

SECONDARY OUTCOMES:
Percent change of Eczema Area and Severity Index (EASI) score from baseline | up to week 18
  The EASI is a composite index with scores ranging from 0 to 72. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) will each be assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe).
Percent change of NRS score from baseline | up to week 18
  The range of Pruritus Numerical Rating Scale (NRS) is from 0 (no itch)-10 (worst imaginable itch)
Body surface area (BSA) of involvement of atopic dermatitis | up to week 18
  Change from baseline in percent of BSA
Children Dermatology Life Quality Index (CDLQI) | up to week 18
  Changes from baseline in CDLQI
Patient-Oriented Eczema Measure (POEM) | up to week 18
  Changes from baseline in POEM
EuroQol Five Dimensions Questionnaire (EQ-5D) | up to week 18
  Changes from baseline in EQ-5D
Safety parameters | up to week 26
  Incidence of Adverse Event(AE), abnormal physical examinations, abnormal vital signs, abnormal ECG, and abnormal lab testing.
Pharmacokinetics parameters | up to week 26
  Trough concentration and exposure of CM310
Pharmacodynamics | up to week 26
  Serum concentration of Thymus and activation regulated chemokine (TARC) , total immunoglobulin E (IgE) and lactate dehydrogenase (LDH)
Immunogenicity | up to week 26
  Detection of anti-drug antibody (ADA)

CONTACTS AND LOCATIONS:
Overall Officials: jianzhong Zhang, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No